CLINICAL TRIAL: NCT00753896
Title: Safety of Exenatide Once Weekly in Patients With Type 2 Diabetes Mellitus Treated With Thiazolidinedione Alone or Thiazolidinedione in Combination With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWDC
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Results first posted 2012-03-20 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: Amylin; Lilly; exenatide once weekly; thiazolidinedione; metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: exenatide — subcutaneous injection, 2.0mcg, once weekly

SUMMARY:
This study will examine the safety of exenatide once weekly (2.0 mg) in approximately 134 patients receiving treatment with thiazolidinedione alone or thiazolidinedione in combination with metformin. Patients are expected to be treated with exenatide once weekly for at least 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes
* At least 18 years of age at screening.
* Have HbA1c of 7.1% to 10.0%, inclusive, at screening.
* Have a body mass index (BMI) of 25 kg/m2 to 45 kg/m2, inclusive.
* Have been treated with a stable dose of TZD (≥4 mg/day rosiglitazone or ≥30 mg/day pioglitazone) for at least 120 days prior to Visit 1 OR Have been treated with a stable dose of TZD (≥4 mg/day rosiglitazone or ≥30 mg/day pioglitazone) for at least 120 days PLUS a stable dose of metformin for at least 90 days prior to Visit 1.
* Have a history of stable body weight (not varying by >10% for at least 3 months prior to screening).
* If female of child-bearing potential (not surgically sterilized and between menarche and 1-year postmenopause) only.

  * Are not breastfeeding.
  * Test negative for pregnancy at the time of screening based on a serum pregnancy test.
  * Intend not to become pregnant during the study.
  * Have practiced a reliable method of birth control (e.g., use of oral contraceptives or approved hormonal implant; diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices; partner with vasectomy; or abstinence) for at least 6 weeks prior to screening.
  * Agree to continue to use a reliable method of birth control (see above) during the study.

Exclusion Criteria:

* Have had a clinically significant history of cardiac disease or presence of active cardiac disease within the year prior to inclusion in the study, including myocardial infarction, clinically significant arrhythmia, unstable angina, coronary artery bypass surgery, angioplasty.
* Is expected to require coronary artery bypass surgery or angioplasty during the course of the study.
* Have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis
* Have a history of renal transplantation or are currently receiving renal dialysis or have serum creatinine ≥135 μmol/L for males and ≥110 μmol/L for females.
* Have active or untreated malignancy, or have been in remission from clinically significant malignancy (other than basal cell or squamous cell skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer) for less than 5 years.
* Have known hemoglobinopathy or chronic anemia (hemoglobin concentration <11.5 g/dL [115 g/L] for males, <10.5 g/dL [105 g/L] for females).
* Have clinically significant history or presence of severe gastrointestinal disease, particularly those which may impact gastric emptying, such as gastroparesis, pyloric stenosis, or gastric bypass surgery.
* Have a history of pancreatitis.
* Have had greater than three episodes of major hypoglycemia within 6 months prior to screening.
* Have any contraindication for the OAD(s) which they use, according to local label requirements.
* Are known to have active proliferative retinopathy.
* Are receiving chronic (>2 weeks) systemic glucocorticoid therapy (excluding topical or inhaled preparations) or have received systemic glucocorticoid therapy for >2 weeks within the 4 weeks immediately preceding screening.
* Have been treated with drugs that promote weight loss (e.g., Xenical® [orlistat], Meridia® [sibutramine], Acomplia® [rimonabant], Acutrim® [phenylpropanolamine], or similar over-the-counter medications) within 3 months of screening.
* Have previously been treated with glucagon-like peptide 1 analogs or liraglutide.
* Have been treated for longer than 2 weeks with any of the following excluded medications within 3 months prior to screening: Insulin; Sulfonylureas; Alpha-glucosidase inhibitors (e.g., Glyset® [miglitol] or Precose® [acarbose]); Meglitinides (e.g., Prandin® [repaglinide] or Starlix® [nateglinide]); Dipeptidyl peptidase (DPP)-4 inhibitors (e.g., Januvia™ [sitagliptin], Galvus® [vildagliptin]); Symlin® (pramlintide acetate).
* Have had an organ transplant.
* Have donated blood within 30 days of screening.
* Have previously completed or withdrawn from this study or any other study investigating exenatide once weekly.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry.
* Are currently participating in an interventional medical, surgical, or pharmaceutical study (a study in which an experimental, drug, medical, or surgical treatment is given). Patients completing the final visit of a study examining safety/efficacy of exenatide BID may enter this study on the same day if they meet other eligibility criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (26):
- United States (11):
  - Research Site, Mesa, Arizona
  - Research Site, Tempe, Arizona
  - Research Site, Concord, California
  - Research Site, Fresno, California
  - Research Site, La Mesa, California
  - Research Site, Atlanta, Georgia
  - Research Site, Idaho Falls, Idaho
  - Research Site, Bowling Green, Kentucky
  - Research Site, Corvallis, Oregon
  - Research Site, Chattanooga, Tennessee
  - Research Site, Memphis, Tennessee
- Canada (4):
  - Research Site, New Westminster, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Cambridge, Ontario
  - Research Site, Windsor, Ontario
- Mexico (3):
  - Research Site, Chihuahua City, Chiuahua
  - Research Site, Monterrey, Nuevo León
  - Research Site, Distrito Federal
- Romania (6):
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Bucharesti
  - Research Site, Craiova
  - Research Site, Iași
  - Research Site, Suceava
- South Africa (2):
  - Research Site, Johannesburg
  - Research Site, Pretoria

REFERENCES:
- [Derived] Norwood P, Liutkus JF, Haber H, Pintilei E, Boardman MK, Trautmann ME. Safety of exenatide once weekly in patients with type 2 diabetes mellitus treated with a thiazolidinedione alone or in combination with metformin for 2 years. Clin Ther. 2012 Oct;34(10):2082-90. doi: 10.1016/j.clinthera.2012.09.007. Epub 2012 Sep 29. PMID 23031623

RESULTS

PARTICIPANT FLOW:
Groups:
- Exenatide Once Weekly: Subcutaneous injection, 2.0mcg, once weekly.
Period: Overall Study
Arm/Group | Exenatide Once Weekly
Started | 134
Completed | 118
Not Completed | 16
Not completed — Adverse Event | 4
Not completed — Death | 1
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — Entry Criteria Not Met | 4

BASELINE CHARACTERISTICS:
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 134
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 114
  >=65 years | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 74
Glycosylated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 7.2 (0.95)
Weight [Mean (Standard Deviation); unit: kg] | 98.1 (18.71)
Background Oral Antidiabetic Agent [Number; unit: participants]
  Metformin + Thiazolidinedione (TZD) | 118
  TZD | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Experiencing Adverse Events
Description: Percentage of patients experiencing treatment-emergent adverse events over 52 weeks
Time Frame: Baseline to Week 52
Population: All enrolled patients who had taken at least one dose of study drug. Sample size based on FDA recommendation for safety exposure: a minimum of 100 patients completing at least 52 weeks of treatment is sought to assess long-term safety associated with exposure to exenatide once weekly.
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 134
percentage of patients | 73.1

2. Primary Outcome: Assessment of Event Rate of Treatment-Emergent Hypoglycemic Events
Description: Major hypoglycemia: any episode with symptoms consistent with hypoglycemia that resulted in loss of consciousness or seizure with prompt recovery in response to administration of glucagon or glucose OR documented hypoglycemia (blood glucose <3.0 mmol/L [54 mg/dL]) and required the assistance of another person. Minor hypoglycemia: any sign or symptom associated with hypoglycemia that is either self-treated by the patient or resolves on its own AND has a concurrent finger stick blood glucose <3.0 mmol/L (54 mg/dL) and not classified as major hypoglycemia. Mean event rate = total number of events for all subjects in a treatment regimen / the total number of subject years of exposure for all subjects in that treatment. Standard error = square root of (total number of events / (subject years of exposure)**2).
Time Frame: Baseline to Week 52
Population: as for outcome 1
Measure: Mean (Standard Error); unit: events per subject-year
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 134
events per subject-year
  Major Hypoglycemia | 0.00 (0.000)
  Minor Hypoglycemia | 0.02 (0.014)

3. Secondary Outcome: Change in HbA1c From Baseline to Week 52
Description: Change in HbA1c from baseline to endpoint
Time Frame: Baseline, Week 52
Population: All enrolled patients who had taken at least one dose of study drug. Last observation carried forward. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Mean (Standard Error); unit: percentage of total hemoglobin
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 132
percentage of total hemoglobin | -0.78 (0.07)

4. Secondary Outcome: Percentage of Patients Achieving HbA1c <=7% at Week 52
Description: Percentage of patients achieving HbA1c <=7% at endpoint (for patients with HbA1c >7% at baseline)
Time Frame: Baseline, Week 52
Population: All enrolled patients who had taken at least one dose of study drug and whose baseline HbA1c was > 7% . Last observation carried forward. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 64
percentage of patients | 68.8

5. Secondary Outcome: Percentage of Patients Achieving HbA1c <=6.5% at Week 52
Description: Percentage of patients achieving HbA1c <=6.5% at endpoint (for patients with HbA1c >6.5% at baseline)
Time Frame: Baseline, Week 52
Population: All enrolled patients who had taken at least one dose of study drug and whose baseline HbA1c was > 6.5%. Last observation carried forward. Only patients with non-missing baseline value and at least one non-missing post-baseline value of the response variable were included in analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 96
percentage of patients | 54.2

6. Secondary Outcome: Change in Fasting Serum Glucose From Baseline to Week 52
Description: Change in fasting serum glucose from baseline to endpoint
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 126
mmol/L | -1.59 (0.21)

7. Secondary Outcome: Change in Body Weight From Baseline to Week 52
Description: Change in body weight from baseline to endpoint
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: kg
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 134
kg | -1.50 (0.45)

8. Secondary Outcome: Change in Total Cholesterol From Baseline to Week 52
Description: Change in Total Cholesterol from baseline to endpoint
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 126
mmol/L | -0.18 (0.08)

9. Secondary Outcome: Change in High-density Lipoprotein (HDL) From Baseline to Week 52
Description: Change in HDL from baseline to endpoint
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 126
mmol/L | 0.04 (0.02)

10. Secondary Outcome: Change in Triglycerides From Baseline to Week 52
Description: Change in Triglycerides from baseline to endpoint
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 126
mmol/L | -0.19 (0.07)

11. Secondary Outcome: Change in Blood Pressure From Baseline to Week 52
Description: Change in Systolic and Diastolic Blood Pressure from baseline to endpoint
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Exenatide Once Weekly
Number analyzed (Participants) | 134
mmHg
  Systolic Blood Pressure | -1.69 (1.12)
  Diastolic Blood Pressure | -0.19 (0.70)

ADVERSE EVENTS:
Arm/Group | Exenatide Once Weekly
Serious Adverse Events (participants affected / at risk) | 9/134
Other Adverse Events (participants affected / at risk) | 67/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=134)
Angina pectoris (Cardiac disorders) | 1
Anorectal cellulitis (Infections and infestations) | 1
Aortic aneurysm (Vascular disorders) | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Calculus urinary (Renal and urinary disorders) | 1
Colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Presyncope (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Exenatide Once Weekly (N=134)
Nausea (Gastrointestinal disorders) | 22
Injection site nodule (General disorders) | 15
Nasopharyngitis (Infections and infestations) | 13
Decreased appetite (Metabolism and nutrition disorders) | 12
Headache (Nervous system disorders) | 12
Upper respiratory tract infection (Infections and infestations) | 10
Vomiting (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 8
Dyspepsia (Gastrointestinal disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 7
Influenza (Infections and infestations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days